CLINICAL TRIAL: NCT02964793
Title: Effects of Serial Plotting on Fundal Height Charts on Identification and Outcomes of Small for Gestational Age Infants
Acronym: HPAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC 14.456
Record Dates: First submitted 2016-10-19; First posted 2016-11-16 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Small for Gestational Age
Keywords: Fetal Growth Restriction; Customised Fetal Weight Reference; Estimated fetal Weight; Symphysis Fundal Height
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention consists in the standardization of current practices. Clinicians in the intervention maternity units will follow a standardized protocol, and will be asked to measure SFH at each antenatal appointment, collect EFW from the 3rd trimester US, report these values on the chart, and monitor fetal growth according to the protocol guidelines
  Interventions: Other: intervention group
- Control group (No Intervention): In the control arm women will benefit from the current routine screening practice for growth failure. The management of pregnancies will remain unchanged. Consultants will be free to monitor growth according to their usual practice. In each maternity unit in the control arm, an information session will be organized on site but its content will be limited to the rational, the objectives of the trial and the study logistics.

INTERVENTIONS:
Other: intervention group — The intervention will include
  1. clinician training sessions, designed to raise awareness of the importance of monitoring for FGR and standardizing SFH measurements
  2. the use of SFH charts and EFW customised charts, built with the same software allowing all information to be recorded on an unique document
  3. the use of the EFW values mentioned on US report, to plot EFW on the customised chart
  4. and explicit recommendations about interpretation of longitudinal values of SFH and EFW measurements. If slopes through consecutive plots are not parallel to either of the predicted centile lines (90th, 50th, 10th) on the chart, and either of the centile lines are 'crossed', fetal biometry by ultrasound scan will be recommended.
  Arms: Intervention group

SUMMARY:
Fetal Growth Restriction (FGR) remains a challenging topic for clinicians, researchers and policy makers, and a central question is how to improve the performance of screening during pregnancy in order to provide appropriate care. The recent recommendations and reporting of French results have raised awareness of the need to improve growth screening in France. Based on the existing literature, the hypothesis is that a greater investment in growth monitoring based on a more rigorous interpretation of information available from routinely implemented clinical assessment and ultrasound will allow for significant gains in detection. The current context provides the opportunity to evaluate the application of a training program for serial plotting of Symphysis Fundal Height (SFH) and Estimated Fetal Weight (EFW) on customised charts. This intervention is consistent with French guidelines which support the monthly measurement of SFH, the use of Customised Fetal Weight Reference (CFWR), in particular for referral US (Ultrasound) examinations, and the longitudinal interpretation of growth. These guidelines were recently restated in the clinical practice recommendations issued by the French College of Obstetricians and Gynecologists.

The intervention tested in the trial will include training of professionals for standardization of SFH measurement, introduction of software, and recommendations for growth interpretation and referral examinations. Expected benefits are an increase in antenatal identification of growth restricted fetuses without an increase in the FP rate. Such a program will allow identified Small for Gestational Age (SGA) fetuses to receive appropriate antenatal care. This intervention could double the detection rate of SGA births from 20 to 40%, corresponding to 32 000 infants nationwide annually for whom antenatal care could be improved.

Main objective: To test the effectiveness of the serial plotting of SFH and EFW measures on customised percentile charts supported by provider training, versus standard antenatal care, to improve the detection of FGR. The aim of the investigators is to double rates of antenatal detection from 20 to 40% among SGA infants, defined as a birthweight under the 10th percentile for GA.

DETAILED DESCRIPTION:
Type of study Randomized cluster trial

Study objectives:

Main objective : To test the effectiveness of the serial plotting of SFH and EFW measures on customised percentile charts supported by provider training, versus standard antenatal care, to improve the detection of FGR. Our aim is to double rates of antenatal detection from 20 to 40% among SGA infants, defined as a birthweight under the 10th percentile for GA.

Secondary objectives: To measure the impact of screening program on:

1. Perinatal outcomes: stillbirths and neonatal morbidity and mortality including the risk of severe growth restriction (less than the 3rd percentile).
2. Rate of false positives and likelihood ratios of screening policies
3. Modes of onset of labor and of delivery
4. Resource use and costs : the number of antenatal visits and referrals for ultrasound examinations and their indications will be evaluated

Primary endpoint

Detection of FGR during pregnancy, defined as:

* The mention of suspected growth restriction in medical charts
* And either at least one referral for additional US for growth monitoring
* And/Or a provider indicated delivery for FGR among SGA births, defined as infants with a birthweight below the 10th centile of French CFWR.

Secondary endpoints

1. Perinatal outcomes: late fetal death, Apgar score<7 at 5 min, pH<7, resuscitation, severe growth restriction (less than the 3rd percentile), admission to a neonatal unit, neonatal convulsions, intra-ventricular hemorrhage, hypoxic-ischemic encephalopathy, death during hospital stay
2. Rate of false positives (equal to 1-specificity), and likelihood ratios of screening policies and their 95% confidence interval. The rate of FP will be defined as suspected FGR among non-SGA births according to the CFWR.
3. Modes of onset of labor and of delivery: labor induction and indications, caesarean section and indications (including pre-labor caesarean and caesarean section after onset of labor), provider indicated delivery before 37 and before 39 weeks GA
4. Resource use and costs : number of antenatal visits, number of referrals for ultrasound examinations and mean number of US per woman, number of umbilical artery Doppler examinations

Inclusion criteria : Singleton pregnancy, Booking before or at 30 weeks GA in the maternity units , Delivery in the participating units Exclusion criteria : Terminations of pregnancy, Known fibroid uterus or uterine congenital malformations, Refusal to participate, Minor patient

HPAG is a cluster randomized trial involving 16 geographically dispersed French maternity units. In the maternity units randomized to the intervention group, a protocol of growth monitoring supported by prior training of healthcare professionals will be implemented for all pregnant women receiving antenatal care in the unit, whatever the GA or medical or obstetrical risk.

The intervention consists only in the standardization of current practices. Clinicians in the intervention maternity units will follow a standardized protocol, and will be asked to measure SFH at each antenatal appointment, collect EFW from the 3rd trimester US, report these values on the chart, and monitor fetal growth according to the protocol guidelines. Practices will remain unchanged in the control group.

After delivery, inclusion and exclusion criteria will be assessed by independent clinical research investigators, probably midwives. All SGA births and non-SGA births according to the French CFWR will be included to answer the main and secondary objectives.

Data collection will be carried out by the referent midwife. Recorded information will include the antenatal care provided, suspicion of FGR, labor and delivery modes, and neonatal outcomes until discharge home. The use of the intervention will also be assessed in the intervention maternity units by recording information on the presence and completeness of customised charts in the medical records.

Sites : 16 French maternity units

Duration : 24 months, including 6 months of inclusions

Number of participants : 10 000 births (625 per maternity unit)

ELIGIBILITY:
Inclusion Criteria:

Mothers will be recruited after delivery if they fulfill the following criteria:

* Have a singleton pregnancy
* book before or at 30 weeks GA in the maternity units
* and deliver in the participating unit

Exclusion Criteria:

* Terminations of pregnancy
* Known fibroid uterus or uterine congenital malformations
* Refusal to participate
* Minor patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate detection of FGR | at birth
  The primary outcome will be the detection rate of FGR among SGA births, measured in each arm, defined as:
  * suspected growth restriction mentioned in medical charts
  * AND at least one referral for additional US for growth monitoring
  * AND/OR a provider indicated delivery for FGR among the total number of SGA births, defined as infants with a birthweight below the 10th centile of French CFWR.

SECONDARY OUTCOMES:
Number of participants presenting the following perinatal outcomes | at birth
  Perinatal outcomes:
  * late fetal death,
  * Apgar score<7 at 5 min,
  * pH<7,
  * resuscitation,
  * severe growth restriction (less than the 3rd percentile),
  * admission after birth,
  * neonatal convulsions,
  * intra-ventricular hemorrhage,
  * hypoxic-ischemic encephalopathy,
  * death during hospital stay
Performances of screening policies | at birth
  * Rate of false positives = equal to 1-specificity = 1 - (True negatives/non-SGA births), where True negatives correspond to non-suspected FGR, and its 95% Confidence Interval
  * PLR (positive likelihood ratios = sensibility / (1 - specificity) and its 95% Confidence Interval
  * NLR (negative likelihood ratios = (1 - sensibility) / specificity and its 95% Confidence Interval
Modes of onset of labor and of delivery | at birth
  Modes of onset of labor and of delivery: labor induction and indications, caesarean section and indications (including pre-labor caesarean and caesarean section after onset of labor), provider indicated delivery before 37 and before 39 GA
Resource use and costs | at birth
  Impact of screening program on resource use and costs is characterized by :
  * number of antenatal visits per woman,
  * number of referrals for ultrasound examinations per woman
  * number of umbilical artery Doppler examinations per woman

CONTACTS AND LOCATIONS:
Overall Officials: Anne Ego, PhD, Principal Investigator — University Hospital, Grenoble
Locations (16):
- France (16):
  - Department of Obstetrics and Gynecology, Bordeaux University Hospital, Bordeaux, Bordeaux
  - Department of Obstetrics and Gynecology, Caen University Hospital, Caen, Caen
  - Department of Obstetrics and Gynecology, Louis Mourier Hospital, Assistance Publique-Paris Hospitals (APHP), Colombes
  - Department of Obstetrics and Gynecology, Grenoble University Hospital, Grenoble
  - Department of Obstetrics, Gynecology, and Neonatal Care, Hôpital Jeanne de Flandre, University of Lille, Lille
  - Department of Obstetrics and Gynecology, North Hospital, Assistance Publique-Marseille Hospitals (APHM), Marseille, Marseille
  - Department of Obstetrics and Gynecology, Cochin Hospital, Assistance Publique-Paris Hospitals (APHP), Port Royal, Paris
  - Department of Obstetrics and Gynecology, Trousseau Hospital, Assistance Publique-Paris Hospitals (APHP), Paris
  - Department of Obstetrics and Gynecology, Robert Debré Hospital, Assistance Publique-Paris Hospitals (APHP), Paris, Paris
  - Department of Obstetrics and Gynecology, Antoine Béclère Hospital, Assistance Publique-Paris Hospitals (APHP), Kremlin-Bicêtre, Paris
  - Department of Obstetrics, Hôpital Poissy-Saint Germain, Versailles-St Quentin University, Poissy
  - Department of Obstetrics and Gynecology, Rouen University Hospital, Rouen
  - Department of Perinatality, Obstetrics and Neonatology, Civil hospice Lyon, Saint-Etienne
  - Department of Obstetrics and Gynecology, Hautepierre Hospital, Strasbourg University Hospital, Strasbourg, Strasbourg
  - Department of Obstetrics and Gynecology, Paule de Viguier Hospital, Toulouse University Hospital, Toulouse
  - Department of Obstetrics and Gynecology, Tours University Hospital,, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ego A, Prunet C, Lebreton E, Blondel B, Kaminski M, Goffinet F, Zeitlin J. [Customized and non-customized French intrauterine growth curves. I - Methodology]. J Gynecol Obstet Biol Reprod (Paris). 2016 Feb;45(2):155-64. doi: 10.1016/j.jgyn.2015.08.009. Epub 2015 Sep 28. French. PMID 26422365
- [Background] Ego A, Prunet C, Blondel B, Kaminski M, Goffinet F, Zeitlin J. [Customized and non-customized French intrauterine growth curves. II - Comparison with existing curves and benefits of customization]. J Gynecol Obstet Biol Reprod (Paris). 2016 Feb;45(2):165-76. doi: 10.1016/j.jgyn.2015.08.008. Epub 2015 Oct 1. French. PMID 26431620
- [Background] Monier I, Blondel B, Ego A, Kaminiski M, Goffinet F, Zeitlin J. Poor effectiveness of antenatal detection of fetal growth restriction and consequences for obstetric management and neonatal outcomes: a French national study. BJOG. 2015 Mar;122(4):518-27. doi: 10.1111/1471-0528.13148. Epub 2014 Oct 27. PMID 25346493
- [Background] Ego A. [Definitions: small for gestational age and intrauterine growth retardation]. J Gynecol Obstet Biol Reprod (Paris). 2013 Dec;42(8):872-94. doi: 10.1016/j.jgyn.2013.09.012. Epub 2013 Nov 7. French. PMID 24210714
- [Background] Ego A, Subtil D, Grange G, Thiebaugeorges O, Senat MV, Vayssiere C, Zeitlin J. Customized versus population-based birth weight standards for identifying growth restricted infants: a French multicenter study. Am J Obstet Gynecol. 2006 Apr;194(4):1042-9. doi: 10.1016/j.ajog.2005.10.816. PMID 16580294